Title: Penicillin De-Labeling in the Pediatric Primary Care Setting; Consent Form

NCT Number: 05010304

# Consent to be part of a Research Study To be conducted at

Children's Medical Center of Dallas and any of its affiliated entities

#### **Key Information about this Study**

Most patients labeled as having a penicillin allergy do not have a real allergy and allergy testing is recommended. The purpose of this research study is to determine whether recommended penicillin testing can be performed in the pediatrician's office. Participants will undergo a telephone screening visit to determine eligibility in the study. Participants who choose to participate in the study will undergo penicillin testing and receive amoxicillin when they come to their pediatrician's visit for their annual well child check exam. This visit will take about 2 hours. Follow up phone calls from the study team will occur at 7-10 days after your doctor's visit and again at 1 year.

The greatest risks of this study include the possibility of a reaction to amoxicillin. The most common reaction is a rash that resolves with oral antihistamines, which out of 100 people occurs in approximately 5-15. Serious reactions such as life-threatening anaphylaxis, which can consist of combinations of symptoms such as rash, difficulty breathing, persistent vomiting or diarrhea, and low blood pressure are rare, occurring in less than 1 patient out of a 1000. You will undergo penicillin testing under the supervision of your primary care provider who is trained to recognize and manage such reactions. The possible benefit of your participating in this study is the accurate diagnosis of whether you have a penicillin allergy and limiting the adverse effects of unnecessary penicillin avoidance.

If you are interested in learning more about this study, please continue to read below.

## Information about this form

#### **Enrolling Children or Incompetent Adults**

If you are providing consent for someone else, for example your child, your next-of-kin or someone for whom you are the legal guardian or are designated as a surrogate decision maker on a medical power of attorney, please note that in the sections that follow, the word "you" refers to the person you are providing consent for.

You may be eligible to take part in a research study. This form gives you important information about the study.

Please take time to review this information carefully. You should talk to the researchers about the study and ask them any questions you have. You may also wish to talk to others (for example, your friends, family, or a doctor) about your participation in this study. If you decide to take part in the study, you will be asked to sign this form. Before you sign this form, be sure you understand what the study is about, including the risks and possible benefits to you.

Please tell the researchers or study staff if you are taking part in another research study.

Your doctor is a research investigator in this study. S/he is interested in both your medical care and the conduct of this research study. At any time, you may discuss your care with another doctor who is not part of this research study. You do not have to take part in any research study offered by your doctor.

<u>Voluntary Participation</u> - You do not have to participate if you don't want to. You may also leave the study at any time. If you decide to stop taking part in this research study, it will not affect your relationship with the UT Southwestern staff or doctors. Whether you participate or not will have no effect on your legal rights or the quality of your health care.

If you are a medical student, fellow, faculty, or staff at the Medical Center, your status will not be affected in any way.

STU2021-0517, Chow, FormE-Consent-Main, NS, 10-06-21

# **General Information – "Who is conducting this research?"**

## **Principal Investigator**

The Principal Investigator (PI) is the researcher directing this study; the PI is responsible for protecting your rights, safety and welfare as a participant in the research. The PI for this study is Timothy Chow, MD, Department of Pediatrics at the University of Texas Southwestern Medical Center.

#### **Funding**

The Allergists' Foundation of the American College of Allergy, Asthma, and Immunology, a non-profit organization that promotes scientific research, is funding this study. This organization is providing money to UTSW so that the researchers can conduct the study.

# Purpose - "Why is this study being done?"

While reported adverse reactions to penicillins are common, most patients with a penicillin allergy label can safely tolerate penicillins. As such, proactive evaluation for penicillin allergy has been recommended. As the majority of people note a penicillin allergy in young childhood, pediatricians are uniquely situated to have a significant impact in reducing the long-term consequences of a penicillin allergy label through penicillin testing. Penicillin testing performed by primary care providers such as pediatricians has been performed in other countries, but has not been done in the United States.

You are asked to participate in this research study of penicillin allergy testing in your pediatrician's office. There are many benefits of correctly diagnosing penicillin allergy, as the majority of patients who had a reaction to penicillin will eventually be able to take it again without reaction. Penicillin testing in the pediatrician's office would reduce barriers for testing and increase access to penicillin allergy evaluation.

The researchers hope to learn if penicillin testing can be performed effectively in your pediatrician's office.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# Information about Study Participants – "Who is participating in this research?"

You are being asked to be a participant in this study because you have a penicillin allergy listed in your electronic medical health record and you see one of the providers at the Children's Health Pediatric Group Medical District clinic for your healthcare.

How many people are expected to take part in this study? This study will enroll approximately 500 study participants.

## Information about Study Procedures – "What will be done if you decide to be in the research?"

While you are taking part in this study, you will be asked to attend approximately 1 visit with the researchers or study staff. You will also have approximately 2 follow up telephone calls.

**Screening** – After you sign this consent to participate, exams, tests, and/or procedures may be done as described below to find out if you can continue in the study; this is called screening. We may be able to use the results of exams, tests, and/or procedures you completed before enrolling in this study. You will be told which results we will obtain and which procedures will not have to be repeated. Many of the procedures are

STU2021-0517, Chow, FormE-Consent-Main, NS, 10-06-21

described below as "**standard care**" and would be done even if you do not take part in this research study. You will be told which ones are for "**research only**".

**Screening Procedures:** Physical examination- the results of the physical examination done as part of your standard care will be used.

The research procedures will add approximately 30 minutes to the length of a routine care visit.

The results of the screening exams, tests, and/or procedures will be reviewed to determine whether you will be allowed to continue in the study. If you are not allowed to continue in the study, the researcher will discuss the reasons with you.

## Study Procedures - as a participant, you will undergo the following procedures:

- Study Visit
  - Medical history and physical exam as part of your routine healthcare maintenance visit
  - o You will receive a small dose of amoxicillin (1 mL) and you will be observed for 10 minutes
  - If you do not have any symptoms, you will be given a larger dose of amoxicillin (4 mL) and observed for 50 minutes. This penicillin testing regimen is standard of care, and we are evaluating if it can be done in your pediatrician's office. This will add approximately 30 minutes to the length of a routine healthcare maintenance visit.
  - During the observation period, your healthcare provider will complete your routine healthcare maintenance visit
  - When the observation period after your second dose of amoxicillin is completed, you will receive any recommended vaccinations that your healthcare provider prescribes.
  - You will then be discharged from the clinic
- Follow up telephone call: you will receive a phone call from a study member 7-10 days after your study visit to see if you developed any reactions after you left the clinic. This should take approximately 5-10 minutes.
- Follow up telephone call: you may receive a phone call from a study member about 10-12 months after your visit to follow up on your drug allergies listed in your health record. This should take approximately 5-10 minutes.

# Risks – "What are the risks of participation in the research?"

## Risks from the specific research procedures (drug(s), interventions, or procedures)

There are risks to taking part in this research study. One risk is that you may have side effects while on the study.

Side effects from this study will usually go away soon after you stop taking the amoxicillin. As you will only receive one full dose of amoxicillin, the risk of side effects should be minimized. In rare cases, side effects can be long lasting or may never go away.

Everyone taking part in the study will be watched carefully for any side effects. However, the study doctors don't know all the side effects that may happen. Be sure to tell your study doctor immediately, about any side effect that you have while taking part in the study.

The following section will describe the risks related to each your participation in this research study. You should talk to your study doctor about any side effects or other problems that you have while taking part in the study.

STU2021-0517, Chow, FormE-Consent-Main, NS, 10-06-21

Side effects can range from mild to serious. Serious side effects are those that may require hospitalization, are life threatening or fatal (could cause death). The frequency that people experience a certain side effect can range from many (likely), few (less likely) or only one or two (rarely).

Risks and side effects related to the amoxicillin include those which are:

#### Less Likely, some may be Serious

In <u>100</u> people, approximately <u>5-15</u> may have:

Rash which resolves with oral antihistamines

#### **Rare and Serious**

In 1000 people, approximately <1 may have:

Anaphylaxis

Treatment of individual acute allergic reactions during the conduct of the study may include antihistamines, epinephrine, b-adrenergic agonists, oxygen. The risks of these common medications include the following

- Antihistamines: drowsiness, dizziness, constipation, stomach upset, blurred vision, dry mouth/nose/throat
- Epinephrine: tachycardia, palpitations, nervousness, sweating, nausea, vomiting, trouble breathing, headache, dizziness, anxiety, tremors, pale skin
- o b-adrenergic agonists: nervousness, shaking, headache, dizziness
- These risks will be minimized by appropriate dosing per guideline management of systemic allergic reactions.

For more information about risks and side effects, ask one of the researchers or study staff.

## Risks to an Embryo, Fetus or Breast-fed Infant

**Females:** If you are part of this study while pregnant or breast-feeding an infant, it is possible that you may expose the unborn child or infant to risks. For that reason, pregnant and breast-feeding females can not participate in the study. If you can become pregnant, a pregnancy test will be done (using a urine sample), and it must be negative before you be a part of this study.

If you do become pregnant during this study, you must tell the researchers immediately.

If your parents or guardian asks, we will tell them the results of your pregnancy test.

#### Are there Risks related to withdrawing from the study?

If you decide to withdraw from this study early, please discuss your decision with the principal investigator. The researcher may ask you to complete study withdrawal procedures at a final telephone visit. There is no risk to you if you do not complete the final withdrawal procedures and you can choose not to participate in them.

#### Are there risks if you also participate in other research studies?

Being in more than one research study at the same time may increase the risk to you. It may also affect the results of the studies. You should not take part in more than one study without approval from the researchers.

#### What if a research-related injury occurs?

The researchers have taken steps to minimize the known or expected risks. However, you may still experience problems or side effects, even though the researchers are careful to avoid them. In the event of a research-related injury or if you experience an adverse reaction, please immediately contact your study doctor.

STU2021-0517, Chow, FormE-Consent-Main, NS, 10-06-21

See the section "Contact Information" for phone numbers and additional information. You may also need to tell your regular doctors.

If you are injured or made sick from taking part in this research study, medical care will be provided. This care may be billed to you or your insurance. We have no plans to give you money if you are injured. The investigator can provide you with more information.

If you sign this form, you do not give up your right to seek additional compensation if you are harmed as a result of being in this study.

## Benefits – "How could you or others benefit from your taking part in this study?"

The possible benefit of your participating in this study is the accurate diagnosis of whether you have a penicillin allergy. This will be done in the familiar environment of your primary provider, as one benefit of this study is that you will not need a referral to see another doctor. If you are determined to not be allergic to penicillin, you would have the benefit of using penicillin antibiotic treatment for future infections and reducing the harms associated with a penicillin-allergy label which include prolonged hospital stays, increased surgical site infections, increased rates of Clostridium Difficile infections, and increased healthcare utilization costs when compared to patients without a penicillin allergy label. There is no guarantee or promise that you will receive any benefit from this study.

# Alternative procedures or course of treatment – "What other options are there to participation in this study?"

There are other options available to you. Your other choices may include 1) getting treatment or care without being in a study, 2) taking part in another study, and 3) getting no treatment

## Payments – Will there be any payments for participation?

There will be no payments for participation.

#### Costs – Will taking part in this study cost anything?

Your health insurance company will be billed for the cost of treatments and procedures that would be done whether or not you took part in this study, such as routine healthcare maintenance visit, amoxicillin challenge, and management of reactions. It is important to understand that some insurance companies do not cover some costs (for example, approved drugs used in a way different from the package instructions). If your insurance company does not cover these treatments or procedures, you will be required to pay for them. Ask the researchers if you have any questions about what it will cost you to take part in this study (for example bills, fees, or other costs related to the research).

# Confidentiality - How will your records be kept confidential?

Information we learn about you in this study will be handled in a confidential manner, within the limits of the law. If we publish the results of the study in a scientific journal or book, we will not identify you. The Institutional Review Board and other groups that have the responsibility of monitoring research may want to see study records which identify you as a subject in this study.

Research policies require that private information about you be protected and this is especially true for your health information. However, the law sometimes allows or requires others to see your information. The information given below describes how your privacy and the confidentiality of your research records will be protected in this study. Medical information collected during this study and the results of any test or procedure that may affect your medical care may be included in your medical record. The information included in your

STU2021-0517, Chow, FormE-Consent-Main, NS, 10-06-21

medical record will be available to health care providers and authorized persons including your insurance company.

Research policies require that private information about you be protected and this is especially true for your health information. However, the law sometimes allows or requires others to see your information. The information given below describes how your privacy and the confidentiality of your research records will be protected in this study. Medical information collected during this study and the results of any test or procedure that may affect your medical care may be included in your medical record. The information included in your medical record will be available to health care providers and authorized persons including your insurance company.

#### What is Protected Health Information (PHI)?

Protected Health Information is information about a person's health that includes information that would make it possible to figure out whose it is. According to the law, you have the right to decide who can see your protected health information. If you choose to take part in this study, you will be giving your permission to the investigators and the research study staff (individuals carrying out the study) to see and use your health information for this research study. In carrying out this research, the health information we will see and use about you will include: your medical history, information that we get from your medical record, information that is collected during your participation in the study including medical and treatment history, information you give us during your participation in the study such as during interviews or from questionnaires, demographic information like your age.

We will get this information by asking you and by looking at your chart at Children's Health.

#### How will your PHI be shared?

Because this is a research study, we will be unable to keep your PHI completely confidential. We may share your health information with people and groups involved in overseeing this research study including:

- the Sponsor, American College of Allergy, Asthma, and Immunology, funding the study. The sponsor includes any people, entities, groups or companies working for or with the sponsor or owned by the sponsor. The sponsor will receive written reports about your participation in the research. The sponsor may look at your health information to assure the quality of the information used in the research.
- the members of the local research team.
- The Institutional Review Board, Human Research Protection Program Office and the Compliance Office of the University of Texas Southwestern Medical Center, and other groups that oversee how research studies are carried out.
- The Research offices at the University of Texas Southwestern Medical Center, Children's Medical Center of Dallas and any of its affiliated entities

If you decide to participate in this study, you will be giving your permission for the groups named above, to collect, use and share your health information. If you choose not to let these groups collect, use and share your health information as explained above, you will not be able to participate in the research study.

Parts of your PHI may be photocopied and sent to a central location or it may be transmitted electronically, such as by e-mail or fax. The groups receiving your health information may not be obligated to keep it private. They may pass information on to other groups or individuals not named here.

#### How will your PHI be protected?

In an effort to protect your privacy, the study staff will use code numbers instead of your name, to identify your health information. Initials and numbers will be used on any photocopies of your study records, and other study materials containing health information that are sent outside of the Children's Health and the University

STU2021-0517, Chow, FormE-Consent-Main, NS, 10-06-21

of Texas Southwestern for review or testing. If the results of this study are reported in medical journals or at meetings, you will not be identified.

# Do you have to allow the use of your health information?

You do not have to allow (authorize) the researchers and other groups to see and share your health information. If you choose not to let the researchers and other groups use your health information, there will be no penalties but you will not be allowed to participate in the study.

After you enroll in this study, you may ask the researchers to stop using your health information at any time. However, you need to say this in writing and send your letter to Timothy Chow, MD at 5323 Harry Hines Blvd, Dallas, Texas 75390-8859. If you tell the researchers to stop using your health information, your participation in the study will end and the study staff will stop collecting new health information from you and about you for this study. However, the study staff will continue to use the health information collected up to the time they receive your letter asking them to stop.

## Can you ask to see the PHI that is collected about you for this study?

The federal rules say that you can see the health information that we collect about you and use in this study. Contact the study staff if you have a need to review your PHI collected for this study. involved.

## How long will your PHI be used?

By signing this form, you agree to let us use and disclose your health information for purposes of the study until the end of the study. This permission to use your personal health information expires when the research ends and all required study monitoring is over.

# Contact Information – Who can you contact if you have questions, concerns, comments or complaints?

If you have questions now, feel free to ask us. If you develop a reaction after leaving the clinic, please contact us using the contact information below. If you have additional questions, concerns, comments or complaints later or you wish to report a problem which may be related to this study please contact:

## **Primary contact:**

Timothy Chow, MD can be reached at 214-456-8490 or at the pager number 972-229-0125. To use the pager, you need to have a touch tone (push button) telephone. Dial the pager number as you would any phone number. When you hear 3 short high pitched beeps, dial in the number where you want the doctor to call you back. Push the # button, hang up and wait for the doctor to return your call.

If primary is not available, contact the pager number 214-822-4829 and ask to speak with Timothy Chow, MD.

The University of Texas Southwestern Medical Center Human Research Protection Program (HRPP) oversees research on human subjects. HRPP and Institutional Review Board (IRB) representatives will answer any questions about your rights as a research subject, and take any concerns, comments or complaints you may wish to offer. You can contact the HRPP by calling the office at 214-648-3060.

STU2021-0517, Chow, FormE-Consent-Main, NS, 10-06-21

### **Research Consent & Authorization Signature Section**

<u>If</u> you agree to participate in this research and agree to the use of your protected health information in this research, sign this section. You will be given a copy of this form to keep. You do not waive any of your legal rights by signing this form.

#### SIGN THIS FORM ONLY IF THE FOLLOWING STATEMENTS ARE TRUE:

- You have read (or been read) the information provided above.
- Your questions have been answered to your satisfaction about the research and about the collection, use and sharing of your protected health information.
- You have freely decided to participate in this research or you are voluntarily giving your consent for another person to participate in this study because you believe this person would want to take part if able to make the decision and you believe it is in this person's best interest.
- You understand that a copy of this signed consent document, information about this study, and the
  results of any test or procedure that may affect your medical care, may be included in your medical
  record. Information in your medical record will be available to health care providers and authorized
  persons including your insurance company.
- You authorize the collection, use and sharing of your protected health information (another person's protected health information) as described in this form.
- If you turn 18 years old after signing this consent form, we will request you to re-sign the consent as an adult if you wish to continue to participate

| Surrogate Signature Section | | | |
|---|---|---|---|
| | | | AM<br>PM |
| Printed Name of Participant | Signature of Participant Giving Assent (If incapable of signing, person obtaining consent should initial here) | Date | Time |
| | | | AM<br>PM |
| Printed Name of Person Giving Consent for Participant (If applicable) | Signature of Person Giving Consent □Parent/□Guardian/□Legally Authorized Representative | Date | Time |
| | | | AM<br>PM |
| Printed Name of Person<br>Obtaining Consent | Signature of Person Obtaining<br>Consent | Date | Time |

# 

Signature of Witness

AM PM

Time

Date

Title of Study: Penicillin De-Labeling in the Pediatric Primary Care Setting

Printed Name of Witness